CLINICAL TRIAL: NCT04269174
Title: The Utility of Biofire Filmarray in Evaluation of Entero Pathogens Triggers in Patients With Chronic Diarrhea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaimaa Mahmoud Abd El-mouez (Other)
Responsible Party: Sponsor-Investigator, Shaimaa Mahmoud Abd El-mouez, Principe investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU The utility of Biofire
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Diarrhoea; Antibiotic Resistant Strain; Polymerase Chain Reaction
Keywords: organic and functiona diarrhoea; pattern; utility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic diarrhea is a common condition and a key symptom in many disorders. It is a major cause of morbidity and mortality worldwide and one of the most common reasons for referral to a gastroenterology clinic.The prevalence varies depending on population and the definition of diarrhea used. It affects approximately 5% of the population at any given point in time, although the exact prevalence is unknown. Diarrhea is associated with 4 pathophysiological mechanisms: osmotic, secretory, exudative and altered motility. It is more useful to classify patients presenting with symptoms of diarrhea according to ''functional'' or ''organic'' characteristics. It is usually difficult to make a reliable differentiation between organic and functional causes in patients with chronic diarrhea based only on history and physical examination .

The standard evaluation of patients with chronic diarrhea that begins with a detailed history, a careful physical examination and then basic diagnostic tests is critical for optimal treatment and prevention. Initially, thought needs to exclude several other possibilities as (a) fecal incontinence masquerading as diarrhea, (b) iatrogenic diarrhea due to drugs, surgery, or therapeutic radiation, (c) chronic infections, and (d) irritable bowel syndrome with diarrhea (IBS-D).

The detection of a broad array of potentially offending agents has traditionally required a combination of microbiologic approaches, including bacterial culture, antigen detection, microscopy, and polymerase chain reaction (PCR). The new multiplex PCR-based panels have several advantages over conventional methods including (i) reduced sample volume requirements, (ii) broad coverage without the need to select specific tests, (iii) enhanced ability to detect coinfections (iv) increased sensitivity and specificity as high as 97-100% and (v) higher throughput.The food and drug administration (FDA) cleared and recommended the use of FilmArray GI panel (BioFire Diagnostics), which targets 22 analytes (bacteria with bacterial toxin, viruses, and parasites)

DETAILED DESCRIPTION:
Investigations:

• Routine laboratory investigation: Complete blood picture and differential WBCs count, liver, kidney function tests, RBG, Na, K, CRP, ESR.

• Microbilogical Investigations:

To ensure that good specimens are provided for examination, it is important to note the following:

* A sterile clean dry container must be used for the collection of fecal samples.
* The specimen should be brought to the lab as soon as possible.
* The specimen container should be clearly labeled with the patient's name, date, and time of passage of the specimen.

A) Conventional methods:

Stool samples will be cultured on Selenite broth then subcultured on blood agar, chocolate agar, MacConkeys agar, Sorbitol MacConkys agar: Xylose Lysine Deoxycholate agar (XLD) ,Sabouraud dextrose agar (SDA), blood agar with 10um/ml ampicillin , Cambylobacter CVA agar plates.

1. Identification of the bacterial organism:

   Pure colonies of isolated microorganisms were identified by:
   * Morphology on agar.
   * Gram stain film was made from the growth to identify morphology of the organism.
   * Biochemical reactions tests.
2. Detection of antibiotic sensitivity pattern according to CLSI 2019 by disc diffusion method
3. Confirmation of results by automated microbial system VITEK 2Compact.

B) Multiplex PCR: for Identification of different causative organisms by Biofire microarray (BioMerieux,France)

ELIGIBILITY:
Inclusion Criteria:

* Patients with diarrhea > 4 weeks

Exclusion Criteria:

* Age below 18 years old and diarhhoea < 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic diarrhea recruited from Al-Rajhi Liver Hospital, Assiut University Hospitals, Assiut, Egypt.
  1. Inclusion criteria:
     Patients with diarrhea > 4 weeks
  2. Exclusion criteria:
  Age below 18 years old and diarhhoea < 4 weeks.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of utility of multiplex PCR in diagnosis of patients with chronic diarrhea. | one year
  The performance of the FilmArray test in the diarrhea for each pathogen on the panel.
To identify antibiotic sensitivity pattern of microbes | one year
  Antibiotic sensitivity patterns for causative microbes.

SECONDARY OUTCOMES:
Epidemiology of infectious causes in chronic diarrhoea | one year
  causes of chronic diarrhoea of enrolled specimens will be evaluated at the end of the study.

REFERENCES:
- [Result] Maharshak N, Ringel Y, Katibian D, Lundqvist A, Sartor RB, Carroll IM, Ringel-Kulka T. Fecal and Mucosa-Associated Intestinal Microbiota in Patients with Diarrhea-Predominant Irritable Bowel Syndrome. Dig Dis Sci. 2018 Jul;63(7):1890-1899. doi: 10.1007/s10620-018-5086-4. Epub 2018 May 17. PMID 29777439
- [Result] Buss SN, Leber A, Chapin K, Fey PD, Bankowski MJ, Jones MK, Rogatcheva M, Kanack KJ, Bourzac KM. Multicenter evaluation of the BioFire FilmArray gastrointestinal panel for etiologic diagnosis of infectious gastroenteritis. J Clin Microbiol. 2015 Mar;53(3):915-25. doi: 10.1128/JCM.02674-14. Epub 2015 Jan 14. PMID 25588652